CLINICAL TRIAL: NCT03212989
Title: IGHID 11627 - A Phase I Study to Evaluate the Effects of Vorinostat and HIV-1 Antigen Expanded Specific T Cell Therapy (HXTC) on Persistent HIV-1 Infection in HIV-Infected Individuals Started on Antiretroviral Therapy (The XTRA Study)
Brief Title: Study to Evaluate Effects of Vorinostat and HXTC on Persistent HIV-1 Infection in HIV-Infected Subjects Started on Antiretroviral Therapy (ART)
Acronym: XTRA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-0468; 1R01HL132791-01 (NIH)
Record Dates: First submitted 2017-06-29; First posted 2017-07-11 (Actual); Results first posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-08

CONDITIONS: HIV-1 Infection
Keywords: HIV; HXTC; Antiretroviral Therapy; HIV-Infected; Vorinostat; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VOR + HXTC arm (Experimental): This is an open label single arm study. All eligible participants receive the following interventions:
  * Step 2 - Single dose of Vorinostat (VOR) 400 mg PO
  * Step 4 - Vorinostat (VOR) 400 mg PO every 72 hrs x 10 doses and 2 HXTC infusions
  * Step 5 - Vorinostat (VOR) 400 mg PO every 72 hrs x 10 doses and 2 HXTC infusions
  Interventions: Drug: Vorinostat; Biological: HXTC

INTERVENTIONS:
Drug: Vorinostat — Participants meeting criteria for Step 1 (exhibit ex-vivo response to VOR) will progress to Step 2 where they will receive a single dose of VOR 400 mg followed by a leukapheresis. If an increase in cell-associated HIV RNA (ca-RNA) is observed in-vivo following the single VOR dose, they will be eligible to donate cells for the manufacture of HXTC (Step 3). Successful manufacturing of the HIV-1 antigen expanded specific T cells will progress participants to combination treatment in Steps 4 and 5. In Steps 4 and Step 5, participants will receive two series of VOR dosing and HXTC infusions, for a total 20 doses of VOR 400 mg and 5 HXTC infusions.
  Other Names: ZOLINZA; MK-0683; SAHA
Biological: HXTC — Participants meeting criteria for Step 1 (exhibit ex-vivo response to VOR) will progress to Step 2 where they will receive a single dose of VOR 400 mg followed by a leukapheresis. If an increase in cell-associated HIV RNA (ca-RNA) is observed in-vivo following the single VOR dose, they will be eligible to donate cells for the manufacture of HXTC (Step 3). Successful manufacturing of the HIV-1 antigen expanded specific T cells will progress participants to combination treatment in Steps 4 and 5. In Steps 4 and Step 5, participants will receive two series of VOR dosing and HXTC infusions, for a total 20 doses of VOR 400 mg and 5 HXTC infusions.
  Other Names: HIV-1 antigen expanded specific T-cell

SUMMARY:
This is a phase I, single-site, study to evaluate the effects of VOR and HIV-1 Antigen Expanded Specific T Cell Therapy (HXTC) on persistent HIV-1 Infection in HIV-infected individuals suppressed on ART. Twelve participants with durable viral suppression will be enrolled and will complete the study. All participants will receive the same treatment and if eligible, will be dosed with HXTC and VOR. Participants will continue their baseline ART regimen throughout the study.

DETAILED DESCRIPTION:
Purpose: This study will test the use of special immune system cells called expanded HIV-specific T Cell (HXTC) Therapy to stimulate the immune system to respond better to HIV. HXTC Therapy will be given in combination with the drug Vorinostat (VOR) which has been shown to stimulate some cells infected with HIV to become active and start making HIV virus. The purpose of this study is to:

1. Evaluate the safety of a series of HXTC infusions in combination with serial doses of VOR and
2. Help scientists evaluate ways of re-activating latent (non-active) HIV virus and determine if the immune system can be made stronger to eliminate the activated HIV virus.

Participants: Men and women living with HIV, ≥ 18 and < 65 years of age, with durable viral suppression for ≥ 24 months as measured on standard HIV RNA assays. Eligible participants must be on stable combination ART (cART) and have a CD4 count ≥ 350 cells/mm3. We plan to enroll up to 12 participants at the University of North Carolina at Chapel Hill (UNC) who complete all 6 Steps of this study.

Procedures (methods):

In Step 1 and prior to initiating the two series of VOR and HXTC combined therapies, all participants will undergo study screening and enrollment where they will be required to: 1. Demonstrate a baseline measurement of the frequency of resting CD4 T cell infection ≥ 0.3 infected cells per million as determined by QVOA, as a further decrease from this low frequency of infection cannot be definitively measured given the quantitative viral outgrowth assay (QVOA) threshold.

Participants with an infectious cells per million (IUPM) measurement > or equal to 0.3 will provide whole blood cells for the manufacture of their HXTC product (Step 3). Successful manufacturing of the HIV-1 antigen expanded specific T cells will progress participants to combination treatment in Steps 4 and 5. In Steps 4 and Step 5, participants will receive two series of VOR dosing and HXTC infusions, for a total 20 doses of VOR 400 mg and 5 HXTC infusions.

In the first series (Step 4), participants will receive VOR 400 mg PO every 72 hours for 10 doses and 2 infusions of HXTC. The first HXTC infusion will be administered six hours after the first dose of VOR (HXTC #1) and the 2nd HXTC infusion (HXTC #2) will occur 6 hours after the 6th dose of VOR.

In the second series in Step 5, participants will receive an additional 10 doses of VOR 400 mg PO every 72 hours and 3 HXTC infusions. The first HXTC infusion in Step 5 (HXTC #3) will occur 6 hours after the 11th dose of VOR (1st dose in Step 5), the 2nd HXTC infusion (HXTC #4) will occur 6 hours after the 16th dose of VOR, and the 3rd HXTC infusion (HXTC #5) will occur 1 - 3 days after the 20th dose of VOR.

If there are insufficient cells manufactured to allow 5 infusions at 1 x 10-8 cells/m-2 dose, the dose will be adjusted to allow 5 infusions at a dose > or equal to 5 x 10-7 cells/m-2 but < 1 x 10-8 cells/m-2 dose.

Following the final HXTC infusion, participants move into Step 6 for a minimum of six additional visits: 21-26. The 2nd leukapheresis will occur at Visit 23 (Week 21), approximately 9 weeks after the last HXTC infusion to evaluate the effect of study treatment on the IUPM by QVOA.

All participants who receive greater than 8 doses of VOR (3200 mg) will be required to enter a study cancer registry where they will be contacted once a year for 5 years after completion of their study participation. The registry was created to monitor participants for the development of future malignancies given concern for genotoxic impact with the use of VOR.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years and < 65 years of age at screening
2. Ability and willingness of participant to give written informed consent. NOTE: Due to the lack of foreseeable benefit to study volunteers, the study will not enroll illiterate or mentally incompetent volunteers.
3. Confirmation of HIV-1 infection HIV infection is defined as documentation by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

   NOTE: The term "licensed" refers to a US FDA-approved kit.

   WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
4. On antiretroviral therapy for at least 24 months and on potent antiretroviral therapy for greater than or equal to 6 months prior to Screening (Visit 1).

   Potent ART is defined by current treatment guidelines and consists of at least 2 nucleoside/nucleotide reverse transcriptase inhibitors plus a non-nucleoside reverse transcriptase inhibitor, integrase inhibitor, or a protease inhibitor without interruption (defined as missing more than 9 total days in the 12 weeks prior to Screening.

   Other potent fully suppressive antiretroviral combinations will be considered on a case-by-case basis. Prior changes in or elimination of medications for easier dosing schedule, intolerance, toxicity, or other reasons are permitted if an alternative suppressive regimen was maintained.
5. Ability and willingness of participant to continue ART throughout the study.
6. Able and willing to adhere to protocol therapy, schedule, and judged adherent to antiretroviral therapy (adherence defined in inclusion criterion 4.)
7. Plasma HIV-1 RNA < 50 copies/mL at two time points in the previous 12 months prior to study screening (one time point can be at screening) and never > or equal to 50 copies/mL on two consecutive time points in the last 24 months.

   NOTE: A single unconfirmed plasma HIV RNA > or equal to 50 copies/mL but < 1000 c/mL is allowed if a subsequent assay was < 50 copies/mL; but none in the 6 months preceding the study screening visit.
8. Plasma HIV-1 RNA < 50 copies/mL at screening
9. CD4+ cell count ≥ 350 cells/mm3 at screening
10. No active HCV infection at or within 90 days of screening.

    Note: No active hepatitis C virus (HCV) defined as negative HCV antibody (HCVAb) or if HCVAb is positive, reflex HCV RNA is negative.
11. No active hepatitis B virus (HBV) infection (measureable HBV DNA or HBV surface antigen-positive (HBVsAg+)) at or within 90 days of screening
12. Women with written documentation of any of the following:

    1. prior hysterectomy OR bilateral oophorectomy (removal of both ovaries)
    2. bilateral tubal ligation or non-surgical permanent sterilization
    3. Women with intact uterus and ovaries who have not had a period for ≥ one year AND have a documented follicle stimulating hormone (FSH) level indicating postmenopausal status.
13. All male study volunteers must agree not to participate in a conception process (e.g. active attempt to impregnate, sperm donation, in vitro fertilization) and, if participating in sexual activity that could lead to pregnancy, the male study volunteer and his female partner must use two reliable methods of contraception (condoms, with or without a spermicidal agent; a diaphragm or cervical cap with spermicide; an intrauterine device (IUD); or hormonal-based contraception) simultaneously while receiving the protocol-specified study products and for 6 weeks after stopping the study products. Participants must use a reliable barrier method of contraception (condom, cervical cap) along with another form of contraception.

    NOTE: For female partners who are receiving ritonavir, estrogen-based contraceptives are not reliable and an alternative method should be suggested.
14. Ability and willingness to provide adequate locator information.
15. Ability and willingness to communicate effectively with study personnel
16. Adequate vascular access for HXTC infusion and leukapheresis.
17. Able to swallow pills without difficulty.
18. Potential participant must have adequate organ function as indicated by the following laboratory values:

System Laboratory Value Hematological Absolute neutrophil count (ANC) ≥1,500 /microliter (mcL) Platelets ≥125,000 / mcL Hemoglobin ≥ 12 g/dL (male) and ≥ 11.0 g/dL (females) System Laboratory Value Coagulation Prothrombin Time (PT) or international normalized ratio (INR) ≤1.1x upper limit of normal (ULN) Chemistry K+ levels within normal limits (WNL) Mg++ levels(footnote 1) WNL Glucose Screening serum glucose ≤ Grade 1 (fasting or non- fasting) Albumin ≥ 3.5 g/dL or ≥ lower limit of normal (LLN) Renal Creatinine clearance determined by the Chronic Kidney Disease Epidemiology Collaboration (CKD-Epi) equation found at: https://www.qxmd.com/calculate/calculator_251/egfr-using-ckd-epi eGFR (epidermal growth factor receptor) > 60 mL/min Hepatic Serum total bilirubin Total bilirubin < 1.1 times the ULN range. If total bilirubin is elevated, direct bilirubin must be < 2 times the ULN range.

NOTE: If participant is on an atazanavir-containing therapy, then a direct bilirubin should be measured instead of the total bilirubin and must be ≤ 1.0 mg/dL.

Aspartate Aminotransferase (AST) (SGOT) and Alanine Transaminase (ALT) (SGPT) < 1.25 X ULN Alkaline Phosphatase < 1.25 X ULN Lipase < 1.1 X ULN

Footnote 1: LLN for Mg++ per the clinical laboratory's normal range used for this study is a grade 1 event per Division of AIDS (DAIDS) Toxicity Table and is allowed for eligibility

ULN = upper limit of normal LLN = lower limit of normal WNL = within normal limits

Exclusion Criteria:

1. Known allergy or sensitivity to components of VOR and its analog or to components in the HXTC product.
2. Women without written documentation of menopause (absence of a period for ≥ one year and FSH level indicating menopause), hysterectomy or bilateral oophorectomy, non-surgical permanent sterilization, or bilateral tubal ligation.
3. Untreated syphilis infection (defined as a positive rapid plasma reagin (RPR) without clear documentation of treatment).

   Note: In cases of untreated syphilis, participant may re-screen following documentation of adequate treatment of syphilis
4. All male participants expecting to father children within the projected duration of the study.
5. Receipt of compounds with Histone Deacetylase (HDAC) inhibitor-like activity, such as valproic acid within 30 days prior to screening.
6. Use of any investigational antiretroviral agents within 30 days prior to screening.
7. If the study PI (or designee) is unable to construct a fully active alternative cART regimen based on previous resistance testing and/or treatment history.
8. Use of the following medications that carry risk of torsade des pointes: amiodarone, arsenic trioxide, astemizole, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide, dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, probucol, procainamide, quinidine, sotalol, sparfloxacin, terfenadine, thioridazine.
9. Use of any of the following within 90 days prior to screening: immunomodulatory, cytokine, or growth stimulating factors such as systemic corticosteroids, cyclosporine, methotrexate, azathioprine, anti-CD25 antibody, interferon (IFN), interleukin-2 (IL-2), coumadin, warfarin, or other Coumadin derivative anticoagulants.
10. Prior use of any HIV immunotherapy or HIV vaccine within 6 months prior to Screening, except for prior HXTC infusions.
11. Received any infusion blood product, immune globulin, or hematopoietic growth factors within 90 days prior to study screening.
12. Pregnancy or breast-feeding.
13. History or other clinical evidence of severe illness, malignancy, immunodeficiency other than HIV, or any other condition that would make the participant unsuitable for the study in the opinion of the investigator (or designee).
14. Use of topical steroids over a total area exceeding 15 cm-2 within 30 days prior to Screening.
15. Treatment for an active AIDS-defining opportunistic infection within 90 days prior to Screening.
16. Any active malignancy that may require chemotherapy or radiation therapy.
17. Compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric illness or a physical illness, e.g., infectious disease. Prisoner recruitment and participation is not permitted.
18. Known psychiatric or substance abuse disorders that would interfere with participant's ability to fully cooperate with the requirements of the trial as assessed by the study investigator (or designee).
19. History or other clinical evidence, as assessed by the study PI (or designee), of significant or unstable cardiac disease (e.g., angina, congestive heart failure, recent myocardial infarction, significant arrhythmia requiring medical or surgical therapy) or clinically significant electrocardiogram (ECG) abnormalities.
20. Unable to have a person available to drive participant home at infusion visits.
21. Participation in another investigational clinical research study (with the exception of an antiretroviral treatment trial that uses FDA approved antiretroviral agents) or use of investigational agents within 30 days prior to screening.

NOTE: Co-enrollment in observational only studies is permitted.

NOTE: Co-enrollment in the AIDS Clinical Trials Group (ACTG) 5332 REPRIEVE study (NCT023442900) and using FDA approved pitavastatin is permitted provided participant enrolled on ACTG 5332 and has taken the study provided medication ≥ 4 months.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Margolis, MD, Principal Investigator — University of North Carolina, Chapel Hill; Cynthia Gay, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gay CL, Hanley PJ, Falcinelli SD, Kuruc JD, Pedersen SM, Kirchherr J, Raines SLM, Motta CM, Lazarski C, Chansky P, Tanna J, Shibli A, Datar A, McCann CD, Sili U, Ke R, Eron JJ, Archin N, Goonetilleke N, Bollard CM, Margolis DM. The Effects of Human Immunodeficiency Virus Type 1 (HIV-1) Antigen-Expanded Specific T-Cell Therapy and Vorinostat on Persistent HIV-1 Infection in People With HIV on Antiretroviral Therapy. J Infect Dis. 2024 Mar 14;229(3):743-752. doi: 10.1093/infdis/jiad423. PMID 38349333

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per study protocol, screening and enrollment occur in Step 1. After establishment of the baseline safety (Visit 1) parameters and qualifying for the study per the Inclusion and Exclusion Criteria, the participant is enrolled (Visit 2) and completes the baseline leukapheresis.
Groups:
- Vorinostat (VOR) + HIV-specific T-cell (HXTC) Arm: This is an open label single arm study. All eligible participants receive the following interventions:
  * Step 2 - Single dose of Vorinostat (VOR) 400 mg PO
  * Step 4 - Vorinostat (VOR) 400 mg PO every 72 hrs x 10 doses and 2 HXTC infusions
  * Step 5 - Vorinostat (VOR) 400 mg PO every 72 hrs x 10 doses and 3 HXTC infusions
  Vorinostat and HXTC: In Steps 4 and Step 5, participants will receive two series of VOR dosing and HXTC infusions, for a total 20 doses of VOR 400 mg and 5 HXTC infusions.
Period: Overall Study
Arm/Group | Vorinostat (VOR) + HIV-specific T-cell (HXTC) Arm
Started | 17
Completed Baseline Leukapheresis | 17
First Intervention Series VOR/HXTC Infusion | 9
Second Intervention Series VOR/HXTC Infusion | 9
Completed | 9
Not Completed | 8
Not completed — Physician Decision | 8

BASELINE CHARACTERISTICS:
Groups:
- Vorinostat (VOR) + HIV-specific T Cell (HXTC) Arm: This is an open label single arm study. All eligible participants receive the following interventions:
  * Step 2 - Single dose of Vorinostat (VOR) 400 mg PO
  * Step 4 - Vorinostat (VOR) 400 mg PO every 72 hrs x 10 doses and 2 HXTC infusions
  * Step 5 - Vorinostat (VOR) 400 mg PO every 72 hrs x 10 doses and 3 HXTC infusions
  Vorinostat and HXTC: In Steps 4 and Step 5, participants will receive two series of VOR dosing and HXTC infusions, for a total 20 doses of VOR 400 mg and 5 HXTC infusions.
Arm/Group | Vorinostat (VOR) + HIV-specific T Cell (HXTC) Arm
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: Year] | 52 [25 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants w/ at Least One ≥ Grade 3 Adverse Event That is Possibly or Definitely Related to Vorinostat (VOR) or HIV-specific T Cell (HXTC)
Description: Safety data will include local and systemic signs and symptoms, laboratory measures of safety/toxicity, and all adverse and serious adverse events. Safety data will be routinely collected throughout the duration of the study.
Time Frame: Up to end of study (weeks 16 through 45)
Measure: Count of Participants; unit: Participants
Groups:
- VOR + HXTC Arm: This is an open label single arm study. All eligible participants receive the following interventions:
  * Step 2 - Single dose of Vorinostat (VOR) 400 mg PO
  * Step 4 - Vorinostat (VOR) 400 mg PO every 72 hrs x 10 doses and 2 HXTC infusions
  * Step 5 - Vorinostat (VOR) 400 mg PO every 72 hrs x 10 doses and 3 HXTC infusions
  Vorinostat and HXTC: In Steps 4 and Step 5, participants will receive two series of VOR dosing and HXTC infusions, for a total 20 doses of VOR 400 mg and 5 HXTC infusions.
Arm/Group | VOR + HXTC Arm
Number analyzed (Participants) | 9
Participants | 0

2. Secondary Outcome: Number of Participants Demonstrating an HIV-specific Immune Response to the Combination of Vorinostat (VOR) and HIV-specific T Cells (HXTC) Therapy as Well as a Change in the Frequency of Latent HIV Infection
Description: The change in ex vivo HIV-specific immune response from baseline was measured by interferon-gamma (IFN-γ) ELISpot throughout the study. Change in the frequency of latent HIV infection from baseline to end of study was measured using a quantitative viral outgrowth assay (QVOA). Participants that exhibited any significant changes in both of these measures were considered to have experienced a positive result.
Time Frame: Up to end of study (weeks 16 through 45)
Measure: Count of Participants; unit: Participants
Arm/Group | VOR + HXTC Arm
Number analyzed (Participants) | 9
Participants | 0

ADVERSE EVENTS:
Time Frame: The Adverse Event (AE) reporting period for each participant began when the participant signed the consent and continued through the 30 days following the End of Study (EOS) visit. Prior to study product administration, any AE that occured was collected as concurrent medical history (pre-existing condition) and not as an AE, unless it was due to a protocol-related procedure (e.g., leukapheresis or large blood collection).
Description: After study entry, any new diagnosis or illnesses that developed, grade ≥3 signs and symptoms, signs and symptoms that were related to Vorinostat (VOR) or HIV-specific T cell (HXTC) therapy, and all signs and symptoms that lead to a change in treatment, regardless of grade were recorded. Systematic assessments included routine clinical examination findings, laboratory, and post-infusion monitoring.
Arm/Group | Vorinostat (VOR) + HIV-specific T-cell (HXTC) Arm
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat (VOR) + HIV-specific T-cell (HXTC) Arm (N=9)
Cardiac flutter (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (10)
Fatigue (General disorders) | 4 (13)
Feeling hot (General disorders) | 1 (1)
Infusion site pain (General disorders) | 1 (1)
Edema peripheral (General disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (2)
Oral candidiasis (Infections and infestations) | 1 (1)
Syphilis (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Citrate toxicity (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Post procedural erythema (Injury, poisoning and procedural complications) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1)
Procedural dizziness (Infections and infestations) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 7 (16)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site bruising (Injury, poisoning and procedural complications) | 2 (2)
Vascular access site pain (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site rupture (Injury, poisoning and procedural complications) | 2 (4)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood cholesterol increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (3)
Blood glucose decreased (Investigations) | 1 (1)
Blood glucose increased (Investigations) | 7 (9)
Blood magnesium decreased (Investigations) | 1 (3)
Blood pressure increased (Investigations) | 7 (32)
Blood sodium increased (Investigations) | 1 (1)
Breath sounds abnormal (Investigations) | 1 (1)
Carbon dioxide decreased (Investigations) | 5 (9)
Glomerular filtration rate decreased (Investigations) | 3 (7)
Lipase increased (Investigations) | 1 (1)
Lymph node palpable (Investigations) | 1 (4)
Protein urine present (Investigations) | 2 (2)
Weight decreased (Investigations) | 1 (2)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 3 (5)
Sciatica (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT03212989/Prot_SAP_000.pdf